CLINICAL TRIAL: NCT02554383
Title: Efficacy of Antibiotics in Children With Acute Sinusitis: Which Subgroups Benefit?
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nader Shaikh (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor-Investigator, Nader Shaikh, Associate Professor of Pediatrics, University of Pittsburgh School of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY20110386; U01AI118506 (NIH)
Record Dates: First submitted 2015-09-08; First posted 2015-09-18 (Estimated); Results first posted 2023-06-08 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Sinusitis; Respiratory Tract Infections
Keywords: pediatrics; antibiotics; placebo
MeSH Terms: conditions — Sinusitis; Respiratory Tract Infections | interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment A (Active Comparator): Amoxicillin-clavulanate (90/6.4 mg/kg/d in 2 divided dosed for 10 days)
  Interventions: Drug: Amoxicillin-clavulanate
- Treatment B (Placebo Comparator): Placebo made to match the study antibiotic will be taken bid orally for 10 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amoxicillin-clavulanate — Amoxicillin-clavulanate (90/6.4 mg/kg/d in 2 divided dosed for 10 days)
  Other Names: Augmentin-Extra strength
  Arms: Treatment A
Drug: Placebo — placebo made to match the study antibiotic given twice a day orally for 10 days
  Arms: Treatment B

SUMMARY:
The objective of this trial is to determine whether certain subgroups of children with acute sinusitis exist in whom antibiotic therapy can be appropriately withheld.

DETAILED DESCRIPTION:
The current clinical practice guideline from the American Academy of Pediatrics for the Diagnosis and Management of Acute Bacterial Sinusitis recommends that the diagnosis of acute sinusitis is made when symptoms of an upper respiratory infection (URI) persist beyond 10 days without showing signs of improvement (persistent presentation), when symptoms appear to worsen (on the 6th to 10th day) after a period of improvement (worsening presentation), or when both high fever and purulent nasal discharge are present concurrently for at least 3 consecutive days (severe presentation). In studies to date, children with persistent and worsening presentations comprise >95% of cases. The investigators preliminary data and the available literature suggest that only a subset of children being diagnosed with acute sinusitis on the basis of current criteria are likely to have bacterial disease. This is not entirely surprising because current criteria rely solely on the duration and the quality of respiratory tract symptoms (which are both common and non-specific). Accordingly, it seems likely that many children currently being diagnosed as having acute sinusitis actually have an uncomplicated upper respiratory infection. This is important because acute sinusitis is one of the most common diagnoses for which antimicrobials are prescribed for children in the United States, accounting for 7.9 million prescriptions annually. A critical need thus exists to establish which subgroups of children currently being diagnosed with acute sinusitis actually benefit from antimicrobial therapy.

The objective of this trial is to determine whether certain subgroups of children with acute sinusitis exist in whom antibiotic therapy can be appropriately withheld. This objective will be achieved by conducting a large, randomized, double-blind, placebo-controlled clinical trial in children 2 to 12 years of age with persistent or worsening presentations of acute sinusitis. Based on the investigators preliminary data, the investigators hypothesize that only certain subgroups of children currently being treated for acute sinusitis actually benefit from antimicrobial therapy. By identifying, in a large placebo-controlled trial, subgroups of children who respectively do and do not benefit from antimicrobial therapy, the investigators will be better able to determine which children should be classified as having acute bacterial sinusitis. Accordingly, the results of this trial may impact not only the treatment guidelines for acute sinusitis but also the diagnostic criteria, and will help ensure that, to the extent possible, antibiotic use is limited to appropriate patients. This, in turn, will maximize the likelihood of achieving optimal outcomes and minimize the risk of promoting antibiotic resistance.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for "persistent" or "worsening" presentations of sinusitis
* Baseline score ≥9 on the Pediatric Rhinosinusitis Symptom Scale

Exclusion Criteria:

* Severe presentation (≥3 days of colored nasal discharge and fever ≥39°C
* Asthma/allergic rhinitis explains symptoms
* Allergy to amoxicillin-clavulanate
* Immotile cilia syndrome
* Cystic fibrosis
* Immunodeficiency
* Parental inability to read/write English or Spanish
* Other concurrent infection (e.g., pneumonia, acute otitis media, streptococcal pharyngitis)
* Systemic toxicity
* Wheezing on exam
* Antibiotic use within 15 days

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 515 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2023-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nader Shaikh, MPH, MD, Principal Investigator — University of Pittsburgh; Ellen R Wald, MD, Principal Investigator — University of Wisconsin, American Family Children's Hospital
Locations (6):
- United States (6):
  - Kentucky Pediatric/Adult Research, Bardstown, Kentucky
  - Cyn3rgy Research, Gresham, Oregon
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - WVU Medicine Pediatric and Adolescent Group Practice, Morgantown, West Virginia
  - American Family Children's Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Shaikh N, Hoberman A, Shope TR, Jeong JH, Kurs-Lasky M, Martin JM, Bhatnagar S, Muniz GB, Block SL, Andrasko M, Lee MC, Rajakumar K, Wald ER. Identifying Children Likely to Benefit From Antibiotics for Acute Sinusitis: A Randomized Clinical Trial. JAMA. 2023 Jul 25;330(4):349-358. doi: 10.1001/jama.2023.10854. PMID 37490085

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Children determined to be eligible for the study and whose parents agreed to participation were randomized to one of two treatments arms. At each site of enrollment, within stratum defined by the presence/absence of colored (yellow or green) nasal discharge, children were randomized 1:1 in blocks of four to receive either twice daily amoxicillin-clavulanate or matching placebo. The analyses of study data were based on the randomized treatment assignment.
Groups:
- Placebo: Placebo made to match the study antibiotic (will be taken bid orally for 10 days)
Period: Overall Study
Arm/Group | Amoxicillin-clavulanate | Placebo
Started (Randomized to the treatment group) | 257 | 258
Completed (Parent completed >=2 diaries Days 2-4 and >= 3 diaries Days 5-11, where Day 1 is day of enrollment) | 234 | 239
Not Completed | 23 | 19
Not completed — Ineligible | 3 | 2
Not completed — Parent completed 0 diaries by Day 4 and 0 diaries Days 5-11 | 8 | 6
Not completed — Parent completed 0 diaries by Day 4 and >=1 diary Days 5-11 | 0 | 2
Not completed — Parent completed >=1 diary by Day 4, but <2 diaries Days 2-4 or <3 diaries Days 5-11 | 12 | 9

BASELINE CHARACTERISTICS:
Population: 515 children underwent randomization; 257 were randomized to the amoxicillin-clavulanate group and 258 to the placebo group. 3 and 2, respectively, were found ineligible after randomization. The remaining 254 and 256 participants, respectively, were the basis for analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Amoxicillin-clavulanate | Placebo | Total
Number analyzed (Participants) | 254 | 256 | 510
Age, Customized [Count of Participants; unit: Participants]
  2 - 5 years | 159 | 165 | 324
  6 - 12 years | 95 | 91 | 186
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114 | 122 | 236
  Male | 140 | 134 | 274
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity was reported by the parent.
  Participants
    Hispanic or Latino | 24 | 34 | 58
    Not Hispanic or Latino | 230 | 222 | 452
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race was reported by the parent.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 5 | 5 | 10
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
    Black or African American | 91 | 88 | 179
    White | 128 | 136 | 264
    More than one race | 24 | 21 | 45
    Unknown or Not Reported | 5 | 6 | 11
Study Site [Count of Participants; unit: Participants] — Participating primary care offices were affiliated with the: (1) Children's Hospital of Pittsburgh, Pittsburgh, PA (2) Children's Hospital of Philadelphia, Philadelphia, PA; (3) Kentucky Pediatric and Adult Research, Bardstown, KY (4) University of Wisconsin, Madison, WI, (5) West Virginia University Children's, Morgantown, WV, and (6) Cyn3rgy Research, Gresham, OR.
  Participants
    Pittsburgh, PA | 196 | 194 | 390
    Philadelphia, PA | 1 | 1 | 2
    Bardstown, KY | 37 | 36 | 73
    Madison, WI | 18 | 20 | 38
    Morgantown, WV | 0 | 2 | 2
    Gresham, OR | 2 | 3 | 5
History of Asthma [Count of Participants; unit: Participants]
  Yes | 46 | 48 | 94
  No | 208 | 208 | 416
History of Allergic Rhinitis [Count of Participants; unit: Participants]
  Yes | 78 | 80 | 158
  No | 176 | 176 | 352
Fever [Count of Participants; unit: Participants] — Fever at any time during the illness
  Participants
    Yes | 120 | 136 | 256
    No | 134 | 120 | 254
Exposure to Other Children [Count of Participants; unit: Participants] — Exposure to other children was defined as exposure to at least 3 children for at least 10 hours per week.
  Participants
    Yes | 200 | 217 | 417
    No | 54 | 39 | 93
Type of Presentation [Count of Participants; unit: Participants] — Persistent was defined as the presence of symptoms for 11 days or longer without improvement. Worsening was defined as a period of improvement followed by worsening symptoms on days 6-10
  Participants
    Persistent | 180 | 173 | 353
    Worsening | 74 | 83 | 157
Pediatric Rhinosinusitis Symptom Scale (PRSS) Score [Count of Participants; unit: Participants] — The Pediatric Rhinosinusitis Symptom Scale (PRSS) is a 8 item scale assessing symptoms of sinusitis. Parents are asked how their child has been doing over the last 24 hours by rating each of 8 symptoms - stuffy nose, runny nose, daytime cough, tiredness, irritability, trouble breathing through the nose, nighttime cough & trouble sleeping - as none, almost none, a little, some, a lot & an extreme amount with respective scores of 0, 1, 2, 3, 4 & 5. The 8 ratings were summed to obtain a PRSS score. Scores ranged from 0-40. Higher scores indicate greater severity.
  Participants
    9 -15 | 39 | 29 | 68
    16 -20 | 43 | 49 | 92
    21 -25 | 62 | 73 | 135
    26 -30 | 65 | 65 | 130
    31 -35 | 34 | 34 | 68
    36 -40 | 11 | 6 | 17
Pathogens Cultured from Nasopharynx [Count of Participants; unit: Participants] — Pathogens cultured were Streptococcus pneumoniae, Haemophilus influenzae, and Moraxella catarrhalis.
  Participants
    Yes | 178 | 185 | 363
    No | 76 | 68 | 144
    Unknown | 0 | 3 | 3
Colored Nasal Discharge [Count of Participants; unit: Participants] — Nasal discharge, either yellow or green, was considered colored.
  Participants
    Yes | 171 | 169 | 340
    No | 83 | 87 | 170

OUTCOME MEASURES:

1. Primary Outcome: The Mean Pediatric Rhinosinusitis Symptom Scale (PRSS) Score Over the First 10 Days of Follow-up According to the Presence of Pathogens in the Nasopharynx at Enrollment
Description: The Pediatric Rhinosinusitis Symptom Scale (PRSS) is a 8 item scale assessing symptoms of sinusitis. Parents are asked how their child has been doing over the last 24 hours by rating each of 8 symptoms - stuffy nose, runny nose, daytime cough, tiredness, irritability, trouble breathing through the nose, nighttime cough & trouble sleeping - as none, almost none, a little, some, a lot & an extreme amount with respective scores of 0, 1, 2, 3, 4 & 5. The 8 ratings were summed to obtain a PRSS score. Scores ranged from 0-40. Higher scores indicate greater severity. The parent completed the scale on Day 1 (enrollment) & electronically on diaries evenings Days 2-11. Pathogens cultured were Streptococcus pneumoniae, Haemophilus influenzae, and Moraxella catarrhalis.
Time Frame: Days 2 to 11
Population: The analysis was intention-to-treat (ITT). The overall number of participants analyzed is equal to the number of children randomized & eligible who had results of a nasopharyngeal culture at enrollment and whose parent completed the PRSS at least once Days 2 to 11. For any given day, the total number analyzed plus the total number without diary data available on that day is equal to the overall number of participants analyzed for the respective Arm/Group.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Amoxicillin-clavulanate | Placebo
Number analyzed (Participants) | 246 | 247
Score on a scale
  Presence of 1 or more pathogens in the nasopharynx at enrollment - Day 2: number analyzed (Participants) | 166 | 177
  Presence of 1 or more pathogens in the nasopharynx at enrollment - Day 2 | 17.3 (7.8) | 18.6 (7.6)
  Presence of 1 or more pathogens in the nasopharynx at enrollment - Day 3: number analyzed (Participants) | 162 | 171
  Presence of 1 or more pathogens in the nasopharynx at enrollment - Day 3 | 13.9 (7.7) | 16.6 (7.5)
  Presence of 1 or more pathogens in the nasopharynx at enrollment - Day 4: number analyzed (Participants) | 167 | 169
  Presence of 1 or more pathogens in the nasopharynx at enrollment - Day 4 | 11.8 (7.9) | 13.9 (7.6)
  Presence of 1 or more pathogens in the nasopharynx at enrollment - Day 5: number analyzed (Participants) | 163 | 169
  Presence of 1 or more pathogens in the nasopharynx at enrollment - Day 5 | 10.1 (7.6) | 12.0 (7.0)
  Presence of 1 or more pathogens in the nasopharynx at enrollment - Day 6: number analyzed (Participants) | 160 | 171
  Presence of 1 or more pathogens in the nasopharynx at enrollment - Day 6 | 8.5 (7.1) | 10.9 (6.9)
  Presence of 1 or more pathogens in the nasopharynx at enrollment - Day 7: number analyzed (Participants) | 166 | 175
  Presence of 1 or more pathogens in the nasopharynx at enrollment - Day 7 | 7.3 (6.7) | 8.9 (6.4)
  Presence of 1 or more pathogens in the nasopharynx at enrollment - Day 8: number analyzed (Participants) | 164 | 174
  Presence of 1 or more pathogens in the nasopharynx at enrollment - Day 8 | 6.4 (6.7) | 8.3 (6.9)
  Presence of 1 or more pathogens in the nasopharynx at enrollment - Day 9: number analyzed (Participants) | 158 | 174
  Presence of 1 or more pathogens in the nasopharynx at enrollment - Day 9 | 4.9 (5.8) | 7.4 (6.6)
  Presence of 1 or more pathogens in the nasopharynx at enrollment - Day 10: number analyzed (Participants) | 149 | 169
  Presence of 1 or more pathogens in the nasopharynx at enrollment - Day 10 | 4.2 (5.4) | 6.0 (5.9)
  Presence of 1 or more pathogens in the nasopharynx at enrollment - Day 11: number analyzed (Participants) | 153 | 157
  Presence of 1 or more pathogens in the nasopharynx at enrollment - Day 11 | 3.7 (5.1) | 5.8 (6.5)
  Absence of 1 or more pathogens in the nasopharynx at enrollment - Day 2: number analyzed (Participants) | 69 | 59
  Absence of 1 or more pathogens in the nasopharynx at enrollment - Day 2 | 19.5 (7.3) | 18.7 (7.2)
  Absence of 1 or more pathogens in the nasopharynx at enrollment - Day 3: number analyzed (Participants) | 67 | 59
  Absence of 1 or more pathogens in the nasopharynx at enrollment - Day 3 | 15.5 (8.1) | 15.5 (7.2)
  Absence of 1 or more pathogens in the nasopharynx at enrollment - Day 4: number analyzed (Participants) | 69 | 59
  Absence of 1 or more pathogens in the nasopharynx at enrollment - Day 4 | 11.9 (7.4) | 12.5 (6.7)
  Absence of 1 or more pathogens in the nasopharynx at enrollment - Day 5: number analyzed (Participants) | 67 | 60
  Absence of 1 or more pathogens in the nasopharynx at enrollment - Day 5 | 10.3 (7.4) | 10.5 (6.7)
  Absence of 1 or more pathogens in the nasopharynx at enrollment - Day 6: number analyzed (Participants) | 69 | 60
  Absence of 1 or more pathogens in the nasopharynx at enrollment - Day 6 | 8.1 (7.1) | 9.4 (7.0)
  Absence of 1 or more pathogens in the nasopharynx at enrollment - Day 7: number analyzed (Participants) | 68 | 59
  Absence of 1 or more pathogens in the nasopharynx at enrollment - Day 7 | 6.9 (6.5) | 8.3 (6.7)
  Absence of 1 or more pathogens in the nasopharynx at enrollment - Day 8: number analyzed (Participants) | 66 | 60
  Absence of 1 or more pathogens in the nasopharynx at enrollment - Day 8 | 6.2 (6.4) | 7.4 (6.8)
  Absence of 1 or more pathogens in the nasopharynx at enrollment - Day 9: number analyzed (Participants) | 67 | 60
  Absence of 1 or more pathogens in the nasopharynx at enrollment - Day 9 | 5.4 (6.1) | 6.3 (6.7)
  Absence of 1 or more pathogens in the nasopharynx at enrollment - Day 10: number analyzed (Participants) | 64 | 57
  Absence of 1 or more pathogens in the nasopharynx at enrollment - Day 10 | 4.9 (5.9) | 5.5 (6.5)
  Absence of 1 or more pathogens in the nasopharynx at enrollment - Day 11: number analyzed (Participants) | 61 | 56
  Absence of 1 or more pathogens in the nasopharynx at enrollment - Day 11 | 4.1 (5.5) | 4.1 (5.3)
Statistical Analysis 1: Comparison: Amoxicillin-clavulanate vs Placebo; Null hypothesis: The effect of treatment with antibiotics does not differ in the subgroups of children defined, respectively, by the presence and by the absence of pathogens in the nasopharynx at enrollment, i.e., there is no significant interaction between treatment and pathogens in the nasopharynx; Test type: Superiority; p = 0.02, Mixed Models Analysis — The interactions (1) between treatment & pathogens and (2) between treatment & colored nasal discharge are tested simultaneously; The p value is adjusted for PRSS score at enrollment, diary day, study site, treatment, pathogens, colored nasal discharge & interaction (2)
Statistical Analysis 2: Comparison: Amoxicillin-clavulanate vs Placebo; Null hypothesis: There is no difference between the treatment groups in the subgroup of children defined by the presence of one or more pathogens in the nasopharynx at enrollment; Test type: Superiority; Difference of least-squares means = -1.95, 95% CI 2-sided [-2.40 to -1.51] — The Amoxicillin-clavulanate group represents the first number in the subtraction and the Placebo group represents the second. The estimates are adjusted for PRSS score at enrollment, diary day and study site
Statistical Analysis 3: Comparison: Amoxicillin-clavulanate vs Placebo; Null hypothesis: There is no difference between the treatment groups in the subgroup of children defined by the absence of one or more pathogens in the nasopharynx at enrollment; Test type: Superiority; Difference of least-squares means = -0.88, 95% CI 2-sided [-1.63 to -0.12] — [estimate comment as in outcome 1, analysis 2]

2. Primary Outcome: The Mean Pediatric Rhinosinusitis Symptom Scale (PRSS) Score Over the First 10 Days of Follow-up According to the Presence of Colored Nasal Discharge at Enrollment
Description: The Pediatric Rhinosinusitis Symptom Scale (PRSS) is a 8 item scale assessing symptoms of sinusitis. Parents are asked how their child has been doing over the last 24 hours by rating each of 8 symptoms - stuffy nose, runny nose, daytime cough, tiredness, irritability, trouble breathing through the nose, nighttime cough & trouble sleeping - as none, almost none, a little, some, a lot & an extreme amount with respective scores of 0, 1, 2, 3, 4 & 5. The 8 ratings were summed to obtain a PRSS score. Scores ranged from 0-40. Higher scores indicate greater severity. The parent completed the scale on Day 1 (enrollment) & electronically on diaries evenings Days 2-11. Nasal discharge, either yellow or green, was considered colored.
Time Frame: Days 2 to 11
Population: The analysis was ITT. The overall number of participants analyzed is equal to the number of children randomized & eligible whose parent completed the PRSS at least once Days 2 to 11. For any given day, the total number analyzed plus the total number without diary data available on that day is equal to the overall number of participants analyzed for the respective Arm/Group.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Amoxicillin-clavulanate | Placebo
Number analyzed (Participants) | 246 | 250
Score on a scale
  Presence of colored nasal discharge at enrollment - Day 2: number analyzed (Participants) | 158 | 161
  Presence of colored nasal discharge at enrollment - Day 2 | 18.6 (7.9) | 19.0 (7.2)
  Presence of colored nasal discharge at enrollment - Day 3: number analyzed (Participants) | 154 | 157
  Presence of colored nasal discharge at enrollment - Day 3 | 14.8 (8.3) | 16.6 (7.1)
  Presence of colored nasal discharge at enrollment - Day 4: number analyzed (Participants) | 163 | 155
  Presence of colored nasal discharge at enrollment - Day 4 | 12.1 (8.1) | 13.7 (7.1)
  Presence of colored nasal discharge at enrollment - Day 5: number analyzed (Participants) | 154 | 155
  Presence of colored nasal discharge at enrollment - Day 5 | 10.8 (7.8) | 11.3 (6.8)
  Presence of colored nasal discharge at enrollment - Day 6: number analyzed (Participants) | 154 | 157
  Presence of colored nasal discharge at enrollment - Day 6 | 8.6 (7.1) | 10.5 (6.8)
  Presence of colored nasal discharge at enrollment - Day 7: number analyzed (Participants) | 156 | 160
  Presence of colored nasal discharge at enrollment - Day 7 | 7.4 (6.8) | 8.8 (6.4)
  Presence of colored nasal discharge at enrollment - Day 8: number analyzed (Participants) | 155 | 160
  Presence of colored nasal discharge at enrollment - Day 8 | 6.4 (6.4) | 8.2 (7.1)
  Presence of colored nasal discharge at enrollment - Day 9: number analyzed (Participants) | 152 | 161
  Presence of colored nasal discharge at enrollment - Day 9 | 5.1 (6.1) | 7.0 (6.7)
  Presence of colored nasal discharge at enrollment - Day 10: number analyzed (Participants) | 146 | 155
  Presence of colored nasal discharge at enrollment - Day 10 | 4.4 (5.5) | 5.7 (5.9)
  Presence of colored nasal discharge at enrollment - Day 11: number analyzed (Participants) | 146 | 144
  Presence of colored nasal discharge at enrollment - Day 11 | 3.7 (5.2) | 5.2 (5.9)
  Absence of colored nasal discharge at enrollment - Day 2: number analyzed (Participants) | 77 | 78
  Absence of colored nasal discharge at enrollment - Day 2 | 16.4 (7.1) | 17.6 (8.3)
  Absence of colored nasal discharge at enrollment - Day 3: number analyzed (Participants) | 75 | 76
  Absence of colored nasal discharge at enrollment - Day 3 | 13.3 (6.8) | 15.6 (7.9)
  Absence of colored nasal discharge at enrollment - Day 4: number analyzed (Participants) | 73 | 76
  Absence of colored nasal discharge at enrollment - Day 4 | 11.1 (7.0) | 12.9 (8.0)
  Absence of colored nasal discharge at enrollment - Day 5: number analyzed (Participants) | 76 | 77
  Absence of colored nasal discharge at enrollment - Day 5 | 9.0 (6.8) | 12.1 (7.1)
  Absence of colored nasal discharge at enrollment - Day 6: number analyzed (Participants) | 75 | 77
  Absence of colored nasal discharge at enrollment - Day 6 | 7.8 (7.1) | 10.5 (7.3)
  Absence of colored nasal discharge at enrollment - Day 7: number analyzed (Participants) | 78 | 77
  Absence of colored nasal discharge at enrollment - Day 7 | 6.7 (6.3) | 8.8 (6.7)
  Absence of colored nasal discharge at enrollment - Day 8: number analyzed (Participants) | 75 | 77
  Absence of colored nasal discharge at enrollment - Day 8 | 6.1 (6.9) | 7.7 (6.5)
  Absence of colored nasal discharge at enrollment - Day 9: number analyzed (Participants) | 73 | 76
  Absence of colored nasal discharge at enrollment - Day 9 | 4.9 (5.5) | 7.3 (6.5)
  Absence of colored nasal discharge at enrollment - Day 10: number analyzed (Participants) | 67 | 74
  Absence of colored nasal discharge at enrollment - Day 10 | 4.5 (5.6) | 6.2 (6.4)
  Absence of colored nasal discharge at enrollment - Day 11: number analyzed (Participants) | 68 | 71
  Absence of colored nasal discharge at enrollment - Day 11 | 4.0 (5.2) | 5.7 (6.9)
Statistical Analysis 1: Comparison: Amoxicillin-clavulanate vs Placebo; Null hypothesis: The effect of treatment with antibiotics does not differ in the subgroups of children defined, respectively, by the presence and by the absence of colored nasal discharge at enrollment, i.e., there is no significant interaction between treatment and colored nasal discharge; Test type: Superiority; p = 0.37, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; The p value is adjusted for PRSS score at enrollment, diary day, study site, treatment, pathogens, colored nasal discharge & interaction (1)
Statistical Analysis 2: Comparison: Amoxicillin-clavulanate vs Placebo; Null hypothesis: There is no difference between the treatment groups in the subgroup of children defined by the presence of colored nasal discharge at enrollment; Test type: Superiority; Difference of least-squares means = -1.62, 95% CI 2-sided [-2.09 to -1.16] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Amoxicillin-clavulanate vs Placebo; Null hypothesis: There is no difference between the treatment groups in the subgroup of children defined by the absence of colored nasal discharge at enrollment; Test type: Superiority; Difference of least-squares means = -1.70, 95% CI 2-sided [-2.38 to -1.03] — [estimate comment as in outcome 1, analysis 2]

3. Secondary Outcome: The Distribution of Children Experiencing Treatment Failure (TF)
Description: The Pediatric Rhinosinusitis Symptom Scale (PRSS) is a 8 item scale assessing symptoms of sinusitis. Parents are asked how their child has been doing over the last 24 hours by rating each of 8 symptoms - stuffy nose, runny nose, daytime cough, tiredness, irritability, trouble breathing through the nose, nighttime cough & trouble sleeping - as none, almost none, a little, some, a lot & an extreme amount with respective scores of 0, 1, 2, 3, 4 & 5. The 8 ratings were summed to obtain a PRSS score. Scores ranged from 0-40. Higher scores indicate greater severity. The parent completed the scale on Day 1 (enrollment), electronically evenings Days 2-11 & at the follow-up visit. If, compared to the Day 1 score, there was >20% increase at any time, decrease <2 on Day 3, <20% decrease on Day 4, <20% decrease on 2 consecutive occasions Days 5-11 or <50% decrease at follow-up, then criterion for treatment failure (TF) was met. Multiple imputation was used when data was insufficient to assess TF.
Time Frame: Day of enrollment to the day of the follow-up visit. The mean length of actual follow-up was 13.4 days. For each child with incomplete follow-up, multiple imputation was used and PRSS scores for the remaining days were imputed.
Population: The analysis was ITT. The number of participants is equal to the number of children randomized & eligible.
Measure: Count of Participants; unit: Participants
Arm/Group | Amoxicillin-clavulanate | Placebo
Number analyzed (Participants) | 254 | 256
Participants
  Experienced failure | 76 | 111
  Did not experience failure | 178 | 145
Statistical Analysis 1: Comparison: Amoxicillin-clavulanate vs Placebo; Null hypothesis: There is no difference between the treatment groups in the proportion of children experiencing treatment failure; Test type: Superiority; p = 0.003, Log-binomial regression; The p-value is adjusted for study site and and presence of colored nasal discharge

4. Secondary Outcome: The Distribution of Children Developing Acute Otitis Media (AOM) Over the First 10 Days of Follow-up
Description: AOM is an infection of the middle ear marked by acute symptoms and a bulging tympanic membrane. Its diagnosis coincided with receipt of a systemic antibiotic. Systemic antibiotics include Amoxicillin, Amoxicillin-clavulanate, Azithromycin, Bacillin L-A, Cefdinir, Clindamycin, Doxycycline, Levofloxacin, Ofloxacin & Sulfamethoxazole-Trimethoprim. Start and stop dates were recorded.
Time Frame: Days 2 to 11, where Day 1 is day of enrollment. The mean number of days of follow-up in this interval was 9.8.
Population: The analysis was ITT. The number of participants is equal to the number of children randomized & eligible with follow-up post-enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Amoxicillin-clavulanate | Placebo
Number analyzed (Participants) | 251 | 256
Participants
  Developed AOM | 0 | 8
  Did not develop AOM | 251 | 248
Statistical Analysis 1: Comparison: Amoxicillin-clavulanate vs Placebo; Null hypothesis: There is no difference between the treatment groups in the proportion of children developing AOM over the first 10 days of follow-up; Test type: Superiority; p = .007, Fisher Exact

5. Secondary Outcome: The Distribution of Children Receiving a Systemic Antibiotic Over the First 10 Days of Follow-up
Description: Systemic antibiotics include Amoxicillin, Amoxicillin-clavulanate, Azithromycin, Bacillin L-A, Cefdinir, Clindamycin, Doxycycline, Levofloxacin, Ofloxacin & Sulfamethoxazole-Trimethoprim. Start and stop dates were recorded. The antibiotic received is exclusive of the study product assigned at enrollment.
Time Frame: Days 2 to 11, where Day 1 is day of enrollment. The mean number of days of follow-up in this interval was 9.8.
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Amoxicillin-clavulanate | Placebo
Number analyzed (Participants) | 251 | 256
Participants
  Received a systemic antibiotic | 34 | 66
  Did not receive a systemic antibiotic | 217 | 190
Statistical Analysis 1: Comparison: Amoxicillin-clavulanate vs Placebo; Null hypothesis: There is no difference between the treatment groups in the proportion of children receiving a systemic antibiotic over the first 10 days of follow-up; Test type: Superiority; p < 0.001, Log-binomial regression; The p-value is adjusted for study site and and presence of colored nasal discharge

6. Secondary Outcome: The Distribution of Children for Whom Diarrhea or Generalized Rash Was Reported
Description: The monitoring of adverse events (AEs), i.e. diarrhea or generalized rash, began on Day 1 (enrollment) and continued through Day 23 (the follow-up visit). Diarrhea was the occurrence of 3 or more watery stools on one day or 2 watery stools on each of 2 consecutive days. Parents recorded in daily diaries, Days 1-11, information regarding the occurrence of diarrhea. Additionally, parents were asked at the follow-up visit if their child had diarrhea while on study product.
Time Frame: Day 1 through Day 23.
Population: The analysis was ITT. The number of participants is equal to the number of children randomized & eligible
Measure: Count of Participants; unit: Participants
Arm/Group | Amoxicillin-clavulanate | Placebo
Number analyzed (Participants) | 254 | 256
Participants
  Diarrhea or rash was reported | 31 | 13
  Neither diarrhea nor rash was reported | 223 | 243
Statistical Analysis 1: Comparison: Amoxicillin-clavulanate vs Placebo; Null hypothesis: There is no difference between the treatment groups in the proportion of children for whom diarrhea or generalized rash was reported; Test type: Superiority; p = 0.004, Log-binomial regression; The p-value is adjusted for study site and presence of colored nasal discharge

7. Secondary Outcome: The Distribution of Children Compliant With Study Medication
Description: Compliance, expressed as a percentage, is the total number of doses taken divided by the total number of expected doses. The child is considered compliant if he/she has received at least 70% of the study medication. The parent completed diaries evenings Days 2-11. The diaries included yes/no questions - (1) did your child take the study medication last night and (2) did your child take the study medication this morning? The total number of doses taken was calculated based on the responses to question (1), and accounted for the dose dispensed at enrollment when enrollment was 1pm or earlier on Day 1. The total of expected doses was determined from the responses to questions (1) and (2), and accounted for scenarios in which the child was taken off the study medication by the clinician. In some cases, due to incomplete diaries the information was insufficient to declare a child either compliant or not compliant.
Time Frame: Days 1 to 11, where Day 1 is day of enrollment
Population: The analysis was ITT. The number of participants is equal to the number of children randomized & eligible with information sufficient to determine compliance.
Measure: Count of Participants; unit: Participants
Arm/Group | Amoxicillin-clavulanate | Placebo
Number analyzed (Participants) | 226 | 234
Participants
  Compliant, i.e., received at least 70% of the the study medication | 212 | 221
  Not compliant, i.e., received less than 70% of study medication | 14 | 13
Statistical Analysis 1: Comparison: Amoxicillin-clavulanate vs Placebo; Null hypothesis: There is no difference between the treatment groups in the proportion of children compliant with study product; Test type: Superiority; p = 0.75, Log-binomial regression; The p-value is adjusted for presence of colored nasal discharge

8. Other Pre Specified Outcome: The Distribution of Children With a Nonsusceptible Pathogen at the Follow-up Visit
Description: The nonsusceptible pathogens considered are penicillin-intermediate and penicillin-resistant Streptococcus pneumoniae (SPN) and ß-lactamase-positive Haemophilus influenzae (NTHi). Susceptibility to penicillin was defined as follows: susceptible as a minimum inhibitory concentration (MIC) of <=0.06 μg/mL; intermediate as an MIC of greater than 0.06 to less than 2 μg/mL; and resistant as an MIC of >=2 μg/mL. A nasopharyngeal specimen for bacterial culture was obtained at the time of the follow-up visit, occurring between study days 11 and 23.
Time Frame: The follow-up visit. The mean number of days from enrollment to the follow-up visit was 13.4.
Population: The analysis was ITT. The number of participants is equal to the number of children randomized & eligible with a nasopharyngeal specimen obtained at the time of the follow-up visit
Measure: Count of Participants; unit: Participants
Arm/Group | Amoxicillin-clavulanate | Placebo
Number analyzed (Participants) | 148 | 152
Participants
  Nonsusceptible pathogen at the follow-up visit | 19 | 18
  No nonsusceptible pathogen at the follow-up visit | 129 | 134
Statistical Analysis 1: Comparison: Amoxicillin-clavulanate vs Placebo; Null hypothesis: There is no difference between the treatment groups in the proportion of children with a nonsusceptible pathogen at the follow-up visit; Test type: Superiority; p = 0.63, Log-binomial regression; The p-value is adjusted for study site and presence of colored nasal discharge

ADVERSE EVENTS:
Time Frame: The monitoring of adverse events (AEs) began on Day 1 (enrollment) and continued through Day 23 (the follow-up visit). All recorded AEs were followed to adequate resolution.
Description: Parents recorded in daily diaries, Days 1-11, information regarding the occurrence of diarrhea. Additionally, parents were asked at the follow-up visit if their child had diarrhea while on study product.
Arm/Group | Amoxicillin-clavulanate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/254 | 0/256
Serious Adverse Events (participants affected / at risk) | 0/254 | 0/256
Other Adverse Events (participants affected / at risk) | 29/254 | 12/256
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amoxicillin-clavulanate (N=254) | Placebo (N=256)
Diarrhea (Gastrointestinal disorders) | 29 (31) | 12 (13) — Diarrhea was the occurrence of 3 or more watery stools on one day or 2 watery stools on each of 2 consecutive days.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-02): https://cdn.clinicaltrials.gov/large-docs/83/NCT02554383/Prot_SAP_000.pdf